CLINICAL TRIAL: NCT07251725
Title: Unravelling the Genetic Basis of Familial Pulmonary Fibrosis: A Next-Generation Sequencing Approach to Fibrogenesis and Surfactant Disorder Genes
Brief Title: GEN-FPF: Genetic Exploration of Familial Pulmonary Fibrosis
Acronym: GEN-FPF
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Ilaria Campo, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: GEN-FPF
Record Dates: First submitted 2025-09-25; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Familial Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — EDTA blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FPF: Familial Pulmonary Fibrosis
- IPF: idiopathic pulmonary fibrosis

SUMMARY:
Pulmonary fibrosis (PF) is a progressive lung disease marked by tissue scarring and impaired breathing. Familial pulmonary fibrosis (FPF) makes up 10-20% of PF cases and shares features with idiopathic PF (IPF), but the genetic causes of FPF are not fully understood.

This study focuses on uncovering the genetic basis of FPF by analyzing families with multiple affected members. It targets genes involved in fibrogenesis and surfactant disorders, as familial cases often appear earlier and progress more rapidly than sporadic ones.

Understanding FPF genetics could:

1. Identify new genetic markers for early diagnosis and prognosis.
2. Improve genetic counseling and preventive strategies for affected families.
3. Reveal therapeutic targets for personalized treatments.
4. Highlight shared molecular pathways between familial and idiopathic PF, potentially benefiting a broader patient group.

In summary, the study aims to deepen our understanding of FPF genetics to improve diagnosis, counseling, and treatment for both familial and idiopathic forms of pulmonary fibrosis.

DETAILED DESCRIPTION:
observational study , longitudinal retrospective

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Familial Pulmonary Fibrosis (FPF):

At least two individuals from the same family (first-degree relatives) diagnosed with pulmonary fibrosis based on clinical, radiological, or histopathological criteria (e.g., HRCT pattern consistent with usual interstitial pneumonia, UIP).

Definite or probable FPF diagnosis, according to international classification criteria and verified family history of disease.

Age:

Adults aged 18 years or older at the time of enrollment.

Informed Consent:

Ability and willingness to provide written informed consent (or consent provided by a legally authorized representative).

Willingness to participate in genetic testing, clinical evaluations, and longitudinal follow-up.

Availability of Family Members:

Affected family members with pulmonary fibrosis willing to provide blood samples and clinical information.

Unaffected first-degree relatives willing to participate in genetic testing and family history documentation.

Idiopathic Pulmonary Fibrosis (IPF) Cohort:

Individuals with a confirmed diagnosis of idiopathic pulmonary fibrosis (IPF) according to ATS/ERS 2018 criteria, enrolled as a comparative (non-familial) cohort.

Exclusion Criteria:

Non-Familial Pulmonary Fibrosis:

Individuals with isolated, sporadic pulmonary fibrosis (without a family history) who are not part of the defined IPF control group.

Other Significant Pulmonary Diseases:

Presence of pulmonary diseases unrelated to fibrosis (e.g., chronic obstructive pulmonary disease, asthma, cystic fibrosis, or active pulmonary infection).

Refusal or Withdrawal of Consent:

Individuals unwilling to provide or maintain informed consent for participation, genetic testing, or long-term data use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals diagnosed with familial pulmonary fibrosis (FPF) and their first-degree relatives (affected and unaffected), as well as a comparison cohort of idiopathic pulmonary fibrosis (IPF) patients.
  Participants will be recruited from two Italian centers:
  SC Pneumologia, Fondazione IRCCS Policlinico San Matteo (Pavia) Azienda Ospedaliero Universitaria Careggi (Florence)
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number and Type of Pathogenic or Likely Pathogenic Variants Identified by Next-Generation Sequencing (NGS) | within 24 months of participant enrollment
  dentification and classification of genetic variants detected in genes associated with familial pulmonary fibrosis (FPF) and surfactant metabolism (e.g., SFTPC, SFTPA2, ABCA3, MUC5B). Variants will be classified according to ACMG guidelines and reported as counts and frequencies in the study population.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No